CLINICAL TRIAL: NCT06026618
Title: Perioperative Management of Preoperative Anemia in Colorectal Cancer. Effect of Intravenous Iron Treatment Within a Patient Blood Management on Colorectal Cancer Surgery
Brief Title: Perioperative Management of Preoperative Anemia in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Other Study IDs: 21/19
Record Dates: First submitted 2023-07-11; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Anemia; Colorectal Cancer
Keywords: Anemia; Colorectal Cancer; Intravenous Iron Therapy; Transfusion; Patient Blood Management
MeSH Terms: conditions — Anemia; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- cohort 1: non-anemic patients (Hb > 13 g/dL)
- cohort 2: mildly anemic patients (Hb 12-13 mg/dL) without criteria for IVI therapy
- cohort 3: patients treated with IVI (Hb < 12mg/dL or Hb 12-13mg/dL with iron deficiency or risk factors for bleeding)

SUMMARY:
Both preoperative anemia (PA) and perioperative blood transfusion can contribute on poorer outcomes after colon cancer surgery. Anemia is known to be associated with a slower recovery after surgery thus often worsening short-term results, and allogenic red blood cells transfusion (ARBT) are known to promote systemic inflammatory response and affect overall and cancer-specific survival.

Patient Blood Management (PBM) systems are an evidence-based multimodal approach focused on safe and rational use of blood products, mainly through a proper PA assessment, a minimization of procedural blood loos and strict transfusion policies. Given the high prevalence of PA in patients with colorectal cancer (CRC), and its association with adverse events, it is expected that PBM implementation in said scenario carries a decrease in complications and an improved survival rate. Available literature to date supports preoperative anaemia screening and restrictive transfusion policies, nevertheless barriers exist that limit the expected implementation of PBM systems in colorectal surgery.

The present study aims to evaluate feasibility of a PBM pathway implementation in a high-volume CRC Surgery Unit based on completion of anemia screening and treatment before surgery and changes of allogenic products use along the years. The objective is to estimate the impact of a proper preoperative optimization with iron intravenous infusion (IVI) on PA measured from changes Hemoglobin (Hb) levels in comparison to those of non-anemic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Colorectal Cancer
* Patients with an indication of elective radical surgery

Exclusion Criteria:

* treatment with red blood cells transfusion before assessment in the PBM Anemia Clinic
* non-iron deficient anemia
* treatment with Sucrose-based IVI or Oral Iron (OI) preparations not strictly controlled by the PBM clinic

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with colorrectal cancer attended at the hospital
Sampling Method: Non-Probability Sample
Enrollment: 1294 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin | Baseline and up to 30 days
  Change in serum hemoglobin concentration between baseline (at the moment of initial colorectal clinic visit) and day of surgery

SECONDARY OUTCOMES:
Total iron dose | up to 30 days
  Total iron dose administered from the first visit until surgery
number of days needed to complete treatment | up to 30 days
  days of treatment before surgery
number of complications related to IVI administration | up to 30 days
  number of complications related to IVI administration

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Sant Joan Despí, CSI, Sant Joan Despí, Barcelona, Spain